CLINICAL TRIAL: NCT05165251
Title: Blood Pressure and Lipids Reduction in High Risk Elderly Patients With Isolated Systolic Hypertension
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Ji-Guang Wang, Director of the Shanghai Institute of Hypertension, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PLENISH
Record Dates: First submitted 2021-12-07; First posted 2021-12-21 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Isolated Systolic Hypertension
Keywords: amlodipine; atorvastatin; blood pressure
MeSH Terms: conditions — Isolated Systolic Hypertension | interventions — Amlodipine; Atorvastatin

STUDY DESIGN:
Intervention Model Description: After screening and run-in period, eligible patients will be randomly assigned into amlodipine/atorvastatin group (amlodipine/atorvastatin 5mg QD) or amlodipine group (amlodipine 5mg QD) or lifestyle intervention only group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Amlodipine/atorvastatin (Experimental): amlodipine/atorvastatin (5mg/10mg QD)
  Interventions: Drug: Amlodipine/Atorvastatin 5 Mg-10 Mg ORAL TABLET
- Amlodipine (Active Comparator): amlodipine (5mg QD)
  Interventions: Drug: Amlodipine 5mg
- Lifestyle intervention (Other)
  Interventions: Other: Lifestyle intervention

INTERVENTIONS:
Drug: Amlodipine/Atorvastatin 5 Mg-10 Mg ORAL TABLET — Amlodipine/Atorvastatin 5 Mg-10 Mg ORAL TABLET QD
  Arms: Amlodipine/atorvastatin
Drug: Amlodipine 5mg — amlodipine 5mg QD
  Arms: Amlodipine
Other: Lifestyle intervention — Lifestyle intervention
  Arms: Lifestyle intervention

SUMMARY:
1. Study name: Blood Pressure and Lipids Reduction in High Risk Elderly Patients with Isolated Systolic Hypertension.
2. Medicine: amlodipine/atorvastatin tablet (5mg/10mg) and amlodipine (5mg).
3. Rationale: Because of its extremely high prevalence in older adults, hypertension is a leading cause of preventable morbidity and mortality. Both SBP and DBP increase linearly up to the fifth or sixth decade of life, after which DBP gradually decreases while SBP continues to rise. Thus, isolated systolic hypertension (ISH) is the predominant form of hypertension in older persons. But there's still no evidence whether elderly ISH patients would benefit from blood pressure and lipid lowering therapy.
4. Objective: To demonstrate that blood pressure and lipid lowering therapy is effective and safe in elderly ISH patients.
5. Study design: This is a 12-month prospective, randomized, active-controlled, apen-label, multi-center study, with three treatment groups: amlodipine/atorvastatin (5mg/10mg tablet); amlodipine (5mg tablet) and lifestyle intervention.
6. Study population: Men or women aged between 65 and 79 years will be screened for hypertension. Eligible patients should be untreated patients with isolated systolic hypertension (clinic systolic blood pressure ≥ 130 and < 150mmHg), and diastolic blood pressure <80 mmHg). Patients should have abilities to understand the study requirements and provide informed consent.
7. Randomization and treatment: After screening period by centers, eligible patients will be randomly divided into 3 groups, taking one pill of amlodipine/atorvastatin (5mg/10mg tablet) or amlodipine (5mg tablet) or lifestyle intervention only.
8. Follow-up: After meeting the inclusion criteria, there will be 2-week screening period. Clinic blood pressure, ambulatory blood pressure, home blood pressure, electrocardiography, concomitant medication records and adverse event records will be collected at randomization period. Then patients will be randomly assigned into amlodipine/atorvastatin group and amlodipine group and lifestyle only group. The treatment will be observed for 12 months. There will be 6 visiting points in the treatment period, which will be the 1st month, 2nd month, 3rd month, 6th month, 9th month and 12th month.
9. Sample size: A total of 480 patients should be enrolled in total.
10. Timeline: After obtaining the approval of Ethics Committee of Ruijin Hospital in October 2021, recruitment will start. Patients enrollment and follow-up will be performed between January 2022 to December 2023.

DETAILED DESCRIPTION:
1. Study name: Blood Pressure and Lipids Reduction in High Risk Elderly Patients with Isolated Systolic Hypertension.
2. Medicine: amlodipine/atorvastatin tablet (5mg/10mg) and amlodipine (5mg).
3. Rationale: Because of its extremely high prevalence in older adults, hypertension is a leading cause of preventable morbidity and mortality. Both SBP and DBP increase linearly up to the fifth or sixth decade of life, after which DBP gradually decreases while SBP continues to rise. Thus, isolated systolic hypertension (ISH) is the predominant form of hypertension in older persons. But there's still no evidence whether elderly ISH patients would benefit from blood pressure and lipid lowering therapy.
4. Objective: to demonstrate that blood pressure and lipid lowering therapy is effective and safe in elderly ISH patients.
5. Study design: This is a 12-month prospective, randomized, active-controlled, apen-label, multi-center study, with three treatment groups: amlodipine/atorvastatin (5mg/10mg tablet); amlodipine (5mg tablet) and lifestyle intervention.
6. Study population: men or women aged between 65 and 79 years will be screened for hypertension. Eligible patients should be untreated patients with isolated systolic hypertension (clinic systolic blood pressure ≥ 130 and < 150mmHg), and diastolic blood pressure <80 mmHg). Patients should have abilities to understand the study requirements and provide informed consent.
7. Randomization and treatment: After screening period by centers, eligible patients will be randomly divided into 3 groups, taking one pill of amlodipine/atorvastatin (5mg/10mg tablet) or amlodipine (5mg tablet) or lifestyle intervention only.
8. Follow up: after meeting the inclusion criteria, there will be 2-week screening period. Clinic blood pressure, ambulatory blood pressure, home blood pressure, electrocardiography, concomitant medication records and adverse event records will be collected at randomization period. Then patients will be randomly assigned into amlodipine/atorvastatin group and amlodipine group and lifestyle only group. The treatment will be observed for 12 months. There will be 6 visiting points in the treatment period, which will be the 1st month, 2nd month, 3rd month, 6th month, 9th month and 12th month.
9. Sample size: A total of 480 patients should be enrolled in total.
10. Timeline: After obtaining the approval of Ethics Committee of Ruijin Hospital in October 2021, recruitment will start. Patients enrollment and follow-up will be performed between January 2022 to December 2023.
11. Organization: The Centre for Epidemiological Studies and Clinical Trials, Ruijin Hospital, Shanghai, China.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65-79;
* Isolated systolic hypertension (office systolic blood pressure (SBP) ≥ 130 and < 150 mmHg and office diastolic blood pressure (DBP) < 80 mmHg) in untreated patients；
* Ability to understand the study requirements and provide informed consent.

Exclusion Criteria:

* Hypersensitivity history to any study drug or similar drug；
* Severe renal insufficiency (eGFR < 30 mL/min/1.73m2);
* Hyperkalemia (serum potassium > 5mmol/L);
* Active liver disease or hepatic insufficiency (AST or ALT > 3 times upper limit of normal);
* History of malignancy over the past 5 years;
* Severe disease patients with life expectancy of < 1 year;
* Previous or current diagnosis of heart failure;
* Stroke or myocardial infarction within 6 months;
* Previous or current atrial fibrillation, frequent ventricular premature beats, supraventricular tachycardia;
* Patients who are receiving other study drugs or study medical devices;
* Pregnant or lactating women;
* Other circumstances that patients are not appropriate for the study upon the investigator's judgment.

Ages: 65 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2022-01-04 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in mean office systolic blood pressure after 12-month treatment from baseline in each group | Baseline and 12 months

SECONDARY OUTCOMES:
Change in mean office diastolic blood pressure after 12-month treatment from baseline in each group | Baseline and 12 months
Difference in control rate of clinic and home blood pressure after 12-month treatment in each group | Baseline and 12 months
Difference in control rate of ambulatory blood pressure after 12-month treatment in each group | Baseline and 12 months
Change in ambulatory (24-h mean, daytime and nighttime) blood pressure after 12-month treatment from baseline in each group | Baseline and 12 months
Change in low-density lipoprotein cholesterol after 12-month treatment from baseline in each group | Baseline and 12 months
Change in clinic, ambulatory and home mean blood pressure after 6-month treatment from baseline in each group | Baseline and 6 months
Difference in control rate of clinic, ambulatory and home blood pressure after 6-month treatment in each group | Baseline and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Institute of Hypertension, Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, China